CLINICAL TRIAL: NCT00873106
Title: Retinal Thickness and Volume Estimates Given by Time Domain and Spectral Optical Coherence Tomography
Status: Completed | Type: Observational
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Birgit Sander, ph.d, Glostrup University Hospital, Copenhagen
Other Study IDs: OCT comparison
Record Dates: First submitted 2009-03-18; First posted 2009-04-01 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Healthy; Diabetic Maculopathy
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Optical coherence tomography — Stratus OCT: fast radial lines 3D OCT-1000: radial 2048 and 3D OCT Cirrus HD OCT: 3D OCT

SUMMARY:
The purpose of the present study is to determine if the retinal thickness estimates of the Stratus OCT, the 3D OCT-1000, and the CirrusHD OCT are comparable in diabetic and in healthy individuals (OCT=Optical Coherence Tomography).

ELIGIBILITY:
Inclusion Criteria:

* diabetic retinopathy in the diabetic group
* healthy retinas in the healthy group

Exclusion Criteria:

* not able to cooperate
* retinal disease other than macular oedema
* severe media opacities (e.g. cataract)
* prior macular laser photocoagulation except for large oedemas

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A group of diabetic and healthy participants
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Retinal thickness and retinal volume from each OCT scan | within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dorte Nellemann Thornit, MD, Principal Investigator — Department of Ophthalmology, Glostrup Hospital, University of Copenhagen, Nordre Ringvej 57, DK-2600 Glostrup, Denmark
Locations (1):
- Department of Ophthalmology, Glostrup Hospital, University of Copenhagen, Nordre Ringvej 57, Glostrup Municipality, Copenhagen, Denmark